CLINICAL TRIAL: NCT07145684
Title: Effectiveness of a Culturally Tailored Medical Nutrition Therapy for African Patients With Type 2 Diabetes: The Objectif Santé Diabète Benin (OSanDiaBé) Trial
Brief Title: Culturally Tailored Nutrition Therapy to Improve Dietary Adherence of Type 2 Diabetes Patients in Benin, Africa
Acronym: OSanDiaBé
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Principal Investigator, Halimatou Alaofe, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00002233; K01TW012422 (NIH)
Record Dates: First submitted 2025-08-11; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Cultural Adaptation; Medical Nutrition Therapy; Dietary Adherence; Africa
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSanDiaBé intervention (Experimental): The Objectif Sante Diabète Bénin (OSanDiaBé) intervention group will participate in four individual home sessions and eight group sessions in the first six months, with no contact between months six and twelve. They will receive the OSanDiaBé resource package, which includes weekly presentations, a workbook, and an Eating Plan based on the 4-A framework of food security.
  Interventions: Behavioral: A culturally tailored medical nutrition therapy
- Individual standard care (No Intervention): The Individual standard care arm will be a wait-list control group who will receive standard care, including blood glucose management and general lifestyle advice, and will access the OSanDiaBe program at the end of the intervention for equitable treatment.

INTERVENTIONS:
Behavioral: A culturally tailored medical nutrition therapy — This MNT intervention combines evidence-based menu plans based on the 4A framework of food security with individual nutrition counseling and group diabetes education.
  Arms: OSanDiaBé intervention

SUMMARY:
The clinical trial aims to assess the effectiveness of the Objectif Santé Diabète Benin (OSanDiaBé), a culturally tailored medical nutrition therapy (MNT), in enhancing diabetes management and nutrition choices. It seeks to answer two main questions:

1. Does the culturally tailored MNT lower HbA1c levels at 12 months compared to usual care?
2. Does it improve dietary behaviors at 12 months compared to usual care?

DETAILED DESCRIPTION:
This study is a 12-month, parallel-group, randomized controlled trial involving individuals diagnosed with type 2 diabetes. Participants will be randomly assigned in a 1:1 ratio to either (1) usual care (wait-list control group) or (2) nutrition counseling with group-based education (intervention group). The intervention group will receive the OSanDiaBé resource package, which includes weekly presentations, a workbook, and an Eating Plan based on the 4-A framework of food security. They will participate in four individual home sessions and eight group sessions in the first six months, with no contact between months six and twelve. The primary outcome will be the change in HbA1c levels, while secondary outcomes will include lipid profile, anthropometric measures, dietary adherence, diabetes self-efficacy, and diabetes-related quality of life. All outcomes will be assessed at baseline, 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria

* outpatient in one of the participating health centers
* be aged between 40 and 65 years old,
* have a confirmed diagnosis of T2D for a year or longer,
* with uncontrolled diabetes (HbA1c >7%)
* able to read and write in French or a support who read and write in French
* self-identify as Beninese (born in Benin or have parents from Benin),
* willing to commit to the study and able to attend weekly meetings
* have family member support for behavioral change
* suitable for general diet and lifestyle advice (i.e., no complex diet needs; suitability determined by the referring healthcare provider)
* be willing to provide informed consent to participate.

Exclusion criteria

* being pregnant, breastfeeding or planning pregnancy,
* participants with type 1 diabetes
* use of medication that might affect weight loss
* planning to travel before the end of the intervention
* have recent cardiovascular complications (e.g., myocardial infarction, stroke, and congestive heart failure),
* currently involved in a similar nutritional educational program (to avoid contamination bias).
* unable to provide consent (e.g., cognitive impairment).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-02 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | HbA1c will be assessed at baseline, 3, 6, and 12 months.
  A hemoglobin A1C (HbA1C) test is a blood test that shows the average level of blood glucose over the past two to three months.

SECONDARY OUTCOMES:
Adherence to dietary recommendations | Dietary adherence will be assessed at baseline, 3, 6, and 12 months.
  Dietary adherence will be assessed using the modified UK Diabetes and Diet Questionnaire (UKDDQ), which consists of 22 items on dietary patterns. Responses indicate food consumption frequency and are coded as follows: A=5 (healthy), B=4 (healthy), C=3 (less healthy), D=2 (less healthy), E=1 (unhealthy), F=0 (unhealthy). Final scores range from 0 to 5, with higher scores indicating better dietary habits.
Weight | Weight will be assessed at baseline, 3, 6, and 12 months.
  Weight will be measured in kilograms to the nearest 0.1 kg with a standard weighing scale (Hana model, China) while ensuring the participants wear light clothing and no shoes.
Height | Height will be assessed at baseline, 3, 6, and 12 months.
  Height will be measured with a stadiometer to the nearest 0.1 cm.
Body mass index | BMI will be assessed at baseline, 3, 6, and 12 months.
  The BMI (Body Mass Index) will be calculated using the formula: weight (kg) divided by height (m) squared. We will use WHO classifications for adult BMI: underweight (under 18.5 kg/m2), normal weight (18.5 to 24.9), overweight (25 to 29.9), and obese (30 or more).
Waist circumference | Waist circumference will be assessed at baseline, 3, 6, and 12 months.
  The waist circumference will be measured at the umbilicus using a non-elastic tape measure while the participant stood upright, recorded in centimeters.
Blood pressure | Blood pressure will be assessed at baseline, 3, 6, and 12 months.
  The blood pressure will be measured with a sphygmomanometer.
Lipid profile | Lipid profile will be assessed at baseline, 3, 6, and 12 months.
  Lipid profile will include triglycerides (TG), low-density lipoprotein cholesterol (LDL-C) and high-density lipoprotein cholesterol (HDL-C).
Behavioral outcomes | Behavioral outcomes will be assessed at baseline, 3, 6, and 12 months.
  We will use the Academy's Evidence-Based Nutrition Practice Guidelines (AEBNPG) for MNT to track behavioral changes in meal planning, food preparation, and physical activity, rating adherence on a scale of 1 (never) to 5 (consistently).

CONTACTS AND LOCATIONS:
Overall Officials: Waliou Amoussa-Hounkpatin, PhD, Principal Investigator — Université d'Abomey-Calavi; Edward Bedric, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Abomey-Calavi, Cotonou, Littoral Department, Benin

IPD SHARING:
Plan to Share IPD: Yes
Data obtained from this study may be shared with qualified researchers who have an academic interest in type 2 diabetes. Any data or samples provided will be coded and will not include any personal health information (PHI). Before sharing the data, the request must receive approval, and all necessary agreements (such as a material transfer agreement) must be in place.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication, and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).